CLINICAL TRIAL: NCT02598141
Title: Comparative Evaluation of Two Techniques for the Treatment of Per-operative Bacteriological Samples Associated With Osteo-articular Sepsis: Grinding (Ultra Turrax) Versus Standard Methods
Brief Title: Grinding Versus Standard Methods for the Treatment of Per-operative Bacteriological Samples Associated With Osteo-articular Sepsis
Acronym: IOAP Turrax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2015/NC-01; 2015-A00720-49 (Other: RCB number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Bacterial Infection
Keywords: Protheses, nails, screws or plates
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Per-op biopsy around material (Other): Patients included in this study require biopsies for suspicion of infected osteo-articular materials (implants, protheses, nails, screw, plates).
  Interventions:
  * Biological sampling grinding
  * Biological sampling with standard procedures
  Interventions: Biological: Biological sampling grinding; Biological: Biological sampling with standard procedures

INTERVENTIONS:
Biological: Biological sampling grinding — One half of the biological material collected during the intervetion (according to standard procedures) will be ground using the Ultra Turrax technique before proceeding with culturing.
Biological: Biological sampling with standard procedures — One half of the biological material collected during the intervetion (according to standard procedures) will be treated according to standard techniques before proceeding with culturing.

SUMMARY:
The main objective of this study was to compare the diagnostic capability (sensitivity and specificity) of standard bacteriological analysis made from one or other of the two sampling processing techniques and perioperative management of samples : the Ultra Turrax method that uses grinding versus the standard method.

DETAILED DESCRIPTION:
The secondary objectives of this study are to:

A. Compare the two techniques in terms of bacterial species identified.

B. Compare the diagnostic capabilities (sensitivity and specificity) of the two sample processing techniques depending on the type of analyzed samples (soft tissue, bone tissue) (subgroup analysis).

C. Compare the diagnostic capabilities (sensitivity and specificity) of the two sample processing techniques depending on the type of joint (subgroup analysis).

D. Compare the diagnostic capabilities (sensitivity and specificity) of the two sample processing techniques depending on the type of implanted materials (prosthesis versus other equipment) (subgroup analysis).

E. Develop a culture collection of bacteria isolated from infection osteo-articular protheses.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be insured or beneficiary of a health insurance plan
* The patient is cared for in the operating theater because of a suspicion of an osteo-articular infection involving any type of material (protheses, screws, plates) and requiring bacteriological sampling
* The patient has not taken any antibiotics within the past 15 days

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The subject presents with an osteo-articulaire infection without material
* Systematic samplings from reversals of aseptic prostheses
* Second intervention for the same patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Presence/absence of an osteo-articular infection according to sample that underwent Ultra Turrax® grinding | Baseline
Presence/absence of an osteo-articular infection according to sample that underwent standard treatment | Baseline

SECONDARY OUTCOMES:
Identification of bacterial species | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Cellier, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Brunaud M, Boutet-Dubois A, Pantel A, Salipante F, Coulomb R, Sotto A, Lavigne JP, Cellier N. Improved Microbiological Diagnosis of Bone and Joint Infections Using Mechanical Bead-Milling Extraction of Bone Specimens with the Ultra-Turrax(R) System. Diagnostics (Basel). 2026 Jan 18;16(2):309. doi: 10.3390/diagnostics16020309. PMID 41594285